CLINICAL TRIAL: NCT07244770
Title: The Effects of Some Antihyperglycemic Drugs on Cognitive Function and Risk of Depression of Diabetic Patients
Acronym: MCI
Status: Recruiting | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Lecturer of clinical pharmacy, Beni-Suef University
Other Study IDs: BeniSuef University Hospital
Record Dates: First submitted 2025-01-09; First posted 2025-11-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: MCI
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SGLT2 I Group: T2DM patients given SGLT2 Is + metformin added to standard of care
  Interventions: Drug: SGLT2 Is+METFORMIN
- DPP4I group: T2DM patients given DPP4Is + metformin added to standard of care
  Interventions: Drug: DPP4 Is+metformin
- Control group: T2DM patients given conventional therapy only
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: SGLT2 Is+METFORMIN — Patients administering SGLT2 Is+metformin added to their treatment for at least the past 12 months
  Other Names: Group 1
  Groups: SGLT2 I Group
Drug: DPP4 Is+metformin — Patients administering DPP4 I+ metformin added to their treatment for at least the past 12 months
  Other Names: Group 2
  Groups: DPP4I group
Drug: Control group — patients administered their standard of care without any changes for the past 6 months
  Other Names: Group 3
  Groups: Control group

SUMMARY:
The study aims to investigate the effects of DPP-4 Is+ metformin versus SGLT2 Is + metformin on the risk of cognitive decline and depression in patients with T2DM.

DETAILED DESCRIPTION:
Older people suffering from Type 2 Diabetes Mellitus possess a major risk for age related cognitive dysfunction and dementia, mainly due to vascular complications.

SGLT2 inhibitors and DPP4 inhibitors are antidiabetic medications, have shown promise not only in glycemic control but also in potentially mitigating cognitive decline and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

-

The study participants should meet the following inclusion criteria:

1. T2DM adult subjects (>55 years old) will be eligible to participate.
2. Patients should be taking SGLT2Is+metformin or DDP4Is + metformin for at least 1 year to be eligible.

Exclusion Criteria:

1- Those with type1 diabetes or ketoacidosis, insulin therapy, end organ failure as chronic renal failure, liver, and heart failure, previous history of pancreatitis, history of Alzheimer's disease or any brain insult, and finally pregnant or lactating females will be excluded from the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients (aged above 55 years)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
MCI | Day 1
  Changes in Montreal Cognitive Assessment (MoCA) score
Depression | Day 1
  Changes in Patient Health Questionnaire-9 (PHQ-9) score

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef Hospital, Banī Suwayf, Egypt